CLINICAL TRIAL: NCT03423342
Title: Safety and Tolerability of the Nutritional Supplement, Nicotinamide Riboside, in Systolic Heart Failure
Brief Title: Nicotinamide Riboside in Systolic Heart Failure
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Kevin O'Brien, Professor, Medicine/Cardiology, University of Washington
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Other
Other Study IDs: STUDY00001830; 1R21HL126209-01 (NIH)
Record Dates: First submitted 2017-04-11; First posted 2018-02-06 (Actual); Results first posted 2022-11-16 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-10

CONDITIONS: Heart Failure, Systolic
Keywords: nicotinamide riboside; Nicotinamide-Adenine Dinucleotide
MeSH Terms: conditions — Heart Failure, Systolic | interventions — nicotinamide-beta-riboside

STUDY DESIGN:
Intervention Model Description: 2:1 randomization to nicotinamide riboside vs. matching placebo
Who Masked: Participant, Care Provider, Investigator
Masking Description: Randomization and dispensing of matching placebo will be performed by Investigational Drug Services at the University of Washington
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nicotinamide Riboside (Experimental): Nicotinamide riboside will be supplied as 250mg capsules, to be administered orally. The initial dose will be 1 capsule twice daily, followed by weekly up-titration by 1 capsule/dose to a final dose of 4 capsules (1000mg) twice daily at the end of Week 4. Participants will be continued on the final dose up to the final follow up visit (week 12). If, at any step, a dose increase is not tolerated, the maximum previously-tolerated dose will be continued through to week 12.
  Interventions: Dietary Supplement: nicotinamide riboside
- Placebo (Placebo Comparator): Matching placebo will be supplied as 250mg capsules, to be administered orally. The initial dose will be 1 capsule twice daily, followed by weekly up-titration by 1 capsule/dose to a final dose of 4 capsules (1000mg) twice daily at the end of Week 4. Participants will be continued on the final dose up to the final follow up visit (week 12). If, at any step, a dose increase is not tolerated, the maximum previously-tolerated dose will be continued through to week 12.
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: nicotinamide riboside — nicotinamide riboside capsule
  Other Names: Niagen
  Arms: Nicotinamide Riboside
Drug: Placebo — matching placebo capsule
  Arms: Placebo

SUMMARY:
Mitochondrial dysfunction has been implicated in heart failure (HF), and is associated with an imbalance in intracellular ratio of reduced nicotinamide-adenine dinucleotide (NADH) to oxidized nicotinamide-adenine dinucleotide (NAD), or the NADH/NAD ratio. In mouse models of HF, we have found that normalization of the NADH/NAD, through supplementation with NAD+ precursors, is associated with improvement in cardiac function. This Study will randomize participants with systolic HF (ejection fraction ≤40%) to treatment with the NAD precursor, nicotinamide riboside (NR) or matching placebo, uptitrated to a final oral dose of 1000mg twice daily, to determine the safety and tolerability of NR in participants with systolic HF.

DETAILED DESCRIPTION:
Aim 1: Determine the safety and tolerability of NR in patients with clinically stable, systolic heart failure (LVEF <40%). To accomplish this Aim:

A) a total of 30 participants with clinically stable, systolic heart failure (LVEF <40%) will undergo 2:1 randomization to NR 250mg PO twice daily or matching placebo B) NR (or matching placebo), will be increased weekly by 250mg/dose (500mg/day) to a final dose of 1000mg PO twice daily. Clinic visits with labs bi-weekly during dose escalation will assess HF symptoms and monitor labs [B-type natriuretic peptide (BNP), complete blood count (CBC), glycosylated hemoglobin, alanine aminotransferase (ALT), creatine kinase (CK), insulin/glucose, uric acid, electrolytes, blood urea nitrogen (BUN) and creatinine (Cr).

C) to ensure intermediate-term safety and tolerability, participants will continue on their maximum tolerated dose (of NR or placebo) through Study Week 12

Aim 2: Determine whether, at the doses employed, NR and NAD are detectable in whole blood.

Aim 3 (Exploratory): Assess the range of potential effect sizes of NR on HF surrogate endpoints using:

A) Six-minute walk tests (6MWTs) at each visit (including Screening) to assess functional capacity B) Echocardiography at Baseline and Week 12 to assess LV systolic function (by real-time, 3D echocardiography) and diastolic function (by integrated Doppler and tissue Doppler imaging)

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 and older with systolic heart failure [left ventricular ejection fraction (LVEF) by standard 2D echocardiography or radionuclide ventriculography of ≤40%] deemed, in the clinical opinion of their treating cardiologist to be non-ischemic or ischemic in origin.
* Clinically stable (no cardiac procedures or hospitalizations for hospitalizations for cardiac causes, including HF, ischemia or arrhythmia) within the previous 3 months
* Ability to undergo study procedures, including scheduled visits, blood draws and six-minute walk test (6MWT)
* Willingness/ability to provide informed consent

Exclusion Criteria:

* Heart failure with preserved ejection fraction (LVEF greater than 40%)
* Heart failure due, in the opinion of their treating cardiologist, to etiologies other than non-ischemic or ischemic. Examples of exclusionary heart failure etiologies include primary valvular disease, or infiltrative or inflammatory cardiomyopathies.
* Cardiac surgery, percutaneous coronary intervention (PCI) or cardiac device implantation within the previous 3 months
* Hospitalizations for cardiovascular causes, including heart failure, chest pain, stroke, transient ischemic attack or arrhythmias within the previous 3 months
* Inability to perform Study visits or procedures (e.g., physical inability to perform 6MWT)
* Unwillingness/inability to provide informed consent
* ALT greater than 3 times the upper limit of normal, hepatic insufficiency or active liver disease
* Recent history of acute gout
* Chronic renal insufficiency with creatinine ≥2.5mg/dL
* Pregnant (or likely to become pregnant) women
* Significant co-morbidity likely to cause death in the 6 month follow-up period
* Significant active history of substance abuse within the previous 5 years
* Current participation in another long-term clinical trial
* History of intolerance to NR precursor compounds, including niacin or nicotinamide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-05-19 (Actual); Primary Completion 2019-04-11 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin D O'Brien, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified, public access database will be made available two years after publication of the primary study results. Data files will be delivered in electronic format, providing meta-data that completely describes the tables, variables and coding. Both the raw data and the primary analysis files will be included. Primary analysis files are a compilation of key variables used to generate the statistical results, to help assure that investigators reach consistent conclusions when analyzing the data to published results. Data, documentation and all other materials will be delivered to NHLBI, as well as a document that fully describes the data, steps taken to de-identify the data, and quality control procedures. A document summarizing data tables and other files that are being delivered and describing the data manipulations applied to the data to assure data anonymity, including an annotated clinical study report providing the database variable names.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 2 years following Study completion

REFERENCES:
- [Derived] Wang DD, Airhart SE, Zhou B, Shireman LM, Jiang S, Melendez Rodriguez C, Kirkpatrick JN, Shen DD, Tian R, O'Brien KD. Safety and Tolerability of Nicotinamide Riboside in Heart Failure With Reduced Ejection Fraction. JACC Basic Transl Sci. 2022 Sep 14;7(12):1183-1196. doi: 10.1016/j.jacbts.2022.06.012. eCollection 2022 Dec. PMID 36644285

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nicotinamide Riboside | Placebo
Started | 20 | 10
Completed | 20 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nicotinamide Riboside | Placebo | Total
Number analyzed (Participants) | 20 | 10 | 30
Age, Continuous [Mean (Full Range); unit: years] | 58 [37 to 81] | 60 [39 to 76] | 59 [37 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 15 | 8 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 19 | 9 | 28
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 17 | 10 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 10 | 30
Sitting Blood Pressure Systolic [Mean (Full Range); unit: mmHg] | 106 [65 to 139] | 106 [96 to 122] | 106 [65 to 139]
Sitting Blood Pressure Diastolic [Mean (Full Range); unit: mmHg] | 67 [45 to 104] | 64 [58 to 68] | 66 [45 to 104]
Heart rate [Mean (Full Range); unit: beats/min] | 67 [42 to 84] | 66 [55 to 80] | 67 [45 to 84]
Weight [Mean (Full Range); unit: kg] | 95 [62 to 141] | 96 [56 to 115] | 95 [56 to 141]
Height [Mean (Full Range); unit: cm] | 170 [104 to 196] | 176 [161 to 188] | 172 [104 to 196]
Smoking: Never [Count of Participants; unit: Participants] | 8 | 4 | 12
Alcohol: Never [Count of Participants; unit: Participants] | 3 | 3 | 6
Non-ischemic heart failure [Count of Participants; unit: Participants] | 13 | 6 | 19
Left ventricular (LV) ejection fraction [LV stroke volume (SV)/LV end-diastolic volume (LVEDV)] [Mean (Full Range); unit: percentage of ejection fraction] | 28 [11 to 40] | 28 [14 to 39] | 28 [11 to 40]
Previous myocardial infarction [Count of Participants; unit: Participants] | 7 | 4 | 11
Previous coronary artery bypass surgery [Count of Participants; unit: Participants] | 2 | 4 | 6
Previous percutaneous coronary intervention [Count of Participants; unit: Participants] | 4 | 1 | 5
History of hypertension [Count of Participants; unit: Participants] | 7 | 2 | 9
History of dyslipidemia [Count of Participants; unit: Participants] | 11 | 6 | 17
History of atherosclerotic disease (coronary, peripheral or carotid) [Count of Participants; unit: Participants] | 8 | 4 | 12
History of atrial fibrillation [Count of Participants; unit: Participants] | 6 | 7 | 13
History of atrial flutter [Count of Participants; unit: Participants] | 0 | 3 | 3
History of diabetes [Count of Participants; unit: Participants] | 8 | 1 | 9
Liver disease [Count of Participants; unit: Participants] | 1 | 0 | 1
Emphysema [Count of Participants; unit: Participants] | 1 | 0 | 1
Serum potassium [Mean (Full Range); unit: mEq/L] | 4.2 [3.4 to 4.8] | 4.3 [3.9 to 4.7] | 4.2 [3.4 to 4.8]
Serum glucose [Mean (Full Range); unit: mg/dL] | 131.7 [73.0 to 364.0] | 114.1 [72.0 to 185.0] | 125.8 [72.0 to 364.0]
Serum creatinine [Mean (Full Range); unit: mg/dL] | 1.1 [0.6 to 2.3] | 1.2 [0.6 to 1.7] | 1.1 [0.6 to 2.3]
Alanine aminotransferase, U/L [Mean (Full Range); unit: U/L] | 19.9 [10.0 to 39.0] | 27.3 [16.0 to 40.0] | 22.4 [10.0 to 40.0]
Body temperature [Mean (Full Range); unit: degrees Celsius] | 37 [36 to 37] | 36 [36 to 37] | 37 [36 to 37]
White blood count [Mean (Full Range); unit: cells x 1000/uL] | 6.8 [3.9 to 10.6] | 6.4 [4.1 to 8.5] | 6.7 [3.9 to 10.6]
Hematocrit [Mean (Full Range); unit: %] | 41 [32 to 46] | 42 [34 to 46] | 41 [32 to 46]
Hemoglobin [Mean (Full Range); unit: g/dL] | 13.5 [10.4 to 15.9] | 13.8 [11.5 to 15.9] | 13.6 [10.4 to 15.9]
Platelet count, thousand/uL [Mean (Full Range); unit: cells x 1000/uL] | 194 [113 to 327] | 194 [144 to 263] | 194 [113 to 327]
Aspartate aminotransferase [Mean (Full Range); unit: U/L] | 19.2 [13.0 to 34.0] | 24.9 [18.0 to 42.0] | 21.1 [13.0 to 42.0]
Insulin resistance (homeostasis model assessment) [Mean (Full Range); unit: units] | 7.0 [0.6 to 41.3] | 4.4 [0.7 to 13.6] | 6.1 [0.6 to 41.3]
Estimated glomerular filtration rate [Mean (Full Range); unit: mL/min/1.73_m2] | 71 [31 to 123] | 67 [30 to 109] | 70 [30 to 123]

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability)
Description: Adverse Events
Time Frame: up to 12 weeks
Population: Total Adverse Events, per participant
Measure: Mean (Full Range); unit: events/participant
Arm/Group | Nicotinamide Riboside | Placebo
Number analyzed (Participants) | 20 | 10
events/participant | 3.1 [0.0 to 9.0] | 3.2 [1.0 to 7.0]

2. Secondary Outcome: On-Trial Change in Whole Blood NAD+ Levels
Description: Between-group comparison of On-Trial Change in Whole Blood NAD+ Levels
Time Frame: Week 12-Week 0
Population: Post enrollment, one of the study participants randomized to NR withdraw before the study drug was dispensed.
Measure: Mean (Standard Error); unit: uM
Arm/Group | Nicotinamide Riboside | Placebo
Number analyzed (Participants) | 19 | 10
uM | 29.0 (3.2) | -0.3 (0.6)
Statistical Analysis 1: Comparison: Nicotinamide Riboside; Test type: Superiority; p < 0.0001, t-test, 2 sided — The updated p-value is calculated and not a threshold for statistical significance; Mean Difference (Net) = 30.2, Standard Error of Mean 3.3

3. Secondary Outcome: Number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment
Description: Incidence of On-Trial Abnormal Laboratory Values and/or Adverse Events that Are Related to Treatment
Time Frame: 16 weeks
Measure: Number; unit: participants
Arm/Group | Nicotinamide Riboside | Placebo
Number analyzed (Participants) | 20 | 10
participants | 0 | 0
Statistical Analysis 1: Comparison: Nicotinamide Riboside vs Placebo; Test type: Superiority; p < 0.05, t-test, 2 sided; Mean Difference (Net) = 0, Standard Error of Mean 0

4. Secondary Outcome: Effect of NR on Change in Mitochondrial Function (Maximal Oxygen Consumption Rate)
Description: Mitochondrial Respiration in Isolated Peripheral Blood Mononuclear Cells by the Seahorse (R) Assay
Time Frame: Week 12 - Week 0
Population: One study subject randomized to NR withdrew post enrollment.
Measure: Mean (Standard Error); unit: pmol/min/1,000,000 cells
Arm/Group | Nicotinamide Riboside | Placebo
Number analyzed (Participants) | 19 | 10
pmol/min/1,000,000 cells | 21 (42) | 2 (23)
Statistical Analysis 1: Comparison: Nicotinamide Riboside vs Placebo; Test type: Superiority; p < 0.05, t-test, 2 sided; Mean Difference (Net) = 19, Standard Error of Mean 48

5. Other Pre Specified Outcome: Exploratory Endpoint: Effect of NR on Functional Capacity
Description: Change in Six Minute Walk Distance
Time Frame: Week 12 - Week 0
Measure: Mean (Standard Error); unit: meters
Arm/Group | Nicotinamide Riboside | Placebo
Number analyzed (Participants) | 17 | 9
meters | 6 (8) | 1 (15)
Statistical Analysis 1: Comparison: Nicotinamide Riboside vs Placebo; Test type: Superiority; p < 0.05, t-test, 2 sided; Mean Difference (Net) = 5, Standard Error of Mean 17

6. Other Pre Specified Outcome: Exploratory Endpoint: Effect of NR on Change in Left Ventricular Systolic Function
Description: Change in Left Ventricular Ejection Fraction by 3D-Transthoracic Echocardiography
Time Frame: Week 12 - Week 0
Population: One study subject randomized to NR withdrew post-enrollment. We were unable to obtain the LVEF for one of the enrolled patient randomized to NR.
Measure: Mean (Standard Error); unit: percentage of ejection fraction
Arm/Group | Nicotinamide Riboside | Placebo
Number analyzed (Participants) | 18 | 10
percentage of ejection fraction | 0.0 (2.2) | 0.3 (2.2)
Statistical Analysis 1: Comparison: Nicotinamide Riboside vs Placebo; Test type: Superiority; p < 0.05, t-test, 2 sided; Mean Difference (Net) = 0.3, Standard Error of Mean 3.1

7. Other Pre Specified Outcome: Exploratory Endpoint: Effect of NR on Left Ventricular Diastolic Function
Description: Tissue Doppler Imaging, e'
Time Frame: Week 12 - Week 0
Measure: Mean (Standard Error); unit: cm/sec
Arm/Group | Nicotinamide Riboside | Placebo
Number analyzed (Participants) | 17 | 9
cm/sec | 0.37 (0.54) | -0.44 (0.39)
Statistical Analysis 1: Comparison: Nicotinamide Riboside vs Placebo; Test type: Superiority; p < 0.05, t-test, 2 sided; Mean Difference (Net) = 0.81, Standard Error of Mean 0.66

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Nicotinamide Riboside | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/20 | 2/10
Other Adverse Events (participants affected / at risk) | 19/20 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nicotinamide Riboside (N=20) | Placebo (N=10)
Myalgia, severe (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Heart failure (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nicotinamide Riboside (N=20) | Placebo (N=10)
Nervous system disorders (Nervous system disorders) | 6 (12) | 5 (5)
Infections and infestations (Infections and infestations) | 6 (12) | 5 (5)
Renal and urinary disorders (Renal and urinary disorders) | 1 (1) | 1 (1)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 5 (6) | 1 (1)
General disorders and administration site conditions (General disorders) | 9 (12) | 4 (5)
Gastrointestinal disorders (Gastrointestinal disorders) | 3 (4) | 2 (3)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 3 (8)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Cardiac disorders (Cardiac disorders) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-01-29): https://cdn.clinicaltrials.gov/large-docs/42/NCT03423342/Prot_002.pdf
  • Statistical Analysis Plan (2022-09-27): https://cdn.clinicaltrials.gov/large-docs/42/NCT03423342/SAP_003.pdf